CLINICAL TRIAL: NCT00465439
Title: Randomized Controlled Trial Examining the Effect of Subcutaneous Xylocaine 2% on the Incidence of Vasovagal Reactions and Pain Intensity During Femoral Artery Sheath Removal.
Brief Title: Safety/Efficacy Study of Local Anesthetic Prior to Femoral Artery Sheath Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: A Cook, Hamilton Health Science
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27071995
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Last update posted 2008-08-22 (Estimated); Status verified 2008-08

CONDITIONS: Syncope, Vasovagal; Pain Intensity
Keywords: femoral artery sheath; vasovagal reaction; pain; perception
MeSH Terms: conditions — Syncope, Vasovagal; Pain | interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Subcutaneous Lidocaine 2% (Xylocaine) without epinephrine — 10 ml subcutaneously
  Other Names: Xylocaine 2% without epinephrine

SUMMARY:
This randomized controlled trial will examine the impact of local anesthetic on the frequency of vasovagal reactions and the patients perception of pain during femoral arterial sheath removal after percutaneous coronary intervention.

DETAILED DESCRIPTION:
Patients undergoing percutaneous coronary intervention(PCI) will be randomized to receive subcutaneous local anesthetic (Lidocaine 2% without epinephrine)or no local prior to removal of femoral arterial sheath. They will be assessed for vasovagal reactions and pain intensity during the sheath removal.The incidence of vasovagal reactions and pain intensity scores will be compared between the groups. 200 patients will be enrolled over the course of 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Percutaneous Coronary Intervention
* Femoral arterial sheath

Exclusion Criteria:

* Less than 18 years old
* Emergency procedure
* Transferred out of heart investigation unit prior to sheath removal
* Radial or brachial sheath
* Closure devise
* Venous sheath insitu
* Intra-aortic balloon pump insitu
* Tranvenous pacing
* Mechanical ventilation
* Cognitive impairment
* Unable to read English
* Lidocaine allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2007-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Incidence of vasovagal reaction during femoral sheath removal | During sheath removal
Pain intensity during femoral sheath removal | During sheath removal

CONTACTS AND LOCATIONS:
Overall Officials: Allison Cook, BScN, Principal Investigator — Hamilton Health Science
Locations (1):
- Hamilton Health Science-Heart Investigation Unit, Hamilton, Ontario, Canada